CLINICAL TRIAL: NCT06778200
Title: The Effects of Practitioner Competency and Its Impact on Client Vocational Outcomes When Obtaining a Psychiatric Rehabilitation Certificate
Brief Title: Effects of Practitioner Competency and Impact on Vocational Outcomes
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Mental Health Association (Other)
Responsible Party: Principal Investigator, Dr. Elizabeth Van Houtte, prinicple investigator, University of Manitoba
Other Study IDs: HS 16092 (H2013:033
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2016-07

CONDITIONS: Competence; Consumer Vocational Outcomes; Consumer Satisfaction
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- client responses: The proposed mixed methods study would collect and examine the following information in order to answer the research questions:
  1) The outcomes of clients receiving services from practitioners enrolled in the PVR certificate program before and during the pursuit of the training. (Quantitative
  Interventions: Other: client interview
- practitioner reflections: The proposed mixed methods study would collect and examine the following information in order to answer the research questions:
  1. The perceived competence levels of each practitioner over the course of the PVR curriculum and the corresponding field supervisor's evaluation of competency level using the RICET (Reflective Ipsative Competency Evaluation Tool) . (Quantitative)
  2. A personal reflection paper from each participant which will describe their learning processes as they complete each competency module. (Qualitative)
  Interventions: Other: practitioner responses

INTERVENTIONS:
Other: client interview — using a data collection form clients voluntarily described services provided by practitioner
  Groups: client responses
Other: practitioner responses — completed reflections after each module completion
  Groups: practitioner reflections

SUMMARY:
The following proposal aims to determine if increasing the competency of mental health practitioners (e.g., social workers, occupational therapists, psychiatric nurses) in the area of vocational rehabilitation (VR) helps their clients to realize the benefits of attaining the goals of working (paid and/or volunteer) and/or formal learning. Specifically, we are seeking to answer the following questions:

1. What is the effect of a vocational rehabilitation curriculum on practitioners' competency to set vocational goals for their clients?
2. What is the effect of a vocational rehabilitation curriculum on vocational outcomes of clients served in community mental health centers in Manitoba during and 1 year after practitioners completion of the curriculum?

DETAILED DESCRIPTION:
This proposal is an evaluation of the competencies developed by community health workers through their participation in a vocational rehabilitation curriculum and the aggregate outcomes (employment, education) on a group of their clients over three time periods (before, during and 1 year after participation of the practitioners in the VR curriculum).

Employment and educational opportunities continue to remain elusive goals for persons with a serious mental illness. Community mental health providers agree that work and education are pivotal factors in the recovery process. However, such goals are rarely set, and rarely achieved by the client or the practitioner. "Among those with the most severe and complex mental health problems and illnesses, unemployment is estimated at between 70 and 90 per cent" (Latimer et al 2006). This is the highest rate among all disabilities.

Supported employment is an evidenced based practice, which has shown promising results by addressing many of the barriers to employment and education.. (Bond, 2004; Corbiere, et al 2005). Organizations that offer employment services strive to assist clients in obtaining and maintaining competitive employment. Yet, many staff are uncomfortable or unfamiliar with the very methods and protocols which have been shown to achieve this goal (Corbiere, et al 2010) In the evaluation of employment outcomes of a supported employment housing agency in New Jersey, team members identified lack of competency in vocational rehabilitation approaches as the biggest barrier to employment goals and outcomes (Van Houtte,(2010). From studies and reports, it seems clear that the main barrier encountered in mental health employment service delivery is lack of a workforce competent in evidence-based practice (Hoge, Morris & Paris 2005; Taylor & Bond, 2011).

A number of panels, consortia, and formal reports have indicated the need to improve the service delivery workforce in the mental health field, issuing various "calls for action" (Coursey et al., 2000; U.S. Surgeon General, 1999; New Freedom Commission on Mental Health, 2003; Hoge, et al., 2007; National Alliance for Mental Illness, 2006). The various bodies have consistently identified providers who uphold recovery-based values and attitudes as a critical factor in service delivery, especially in the vocational arena.

Canada's Mental Health Commission (CMHC) recently released 'The Mental Health Strategy of Canada - Changing Directions Changing Lives" (2012). The report specifically addresses rates of employment and human resources development. For example, strategic direction #3 from the CMHC document is to increase the rates of employment for people with mental illness. The recommendations for action 3.5 from the same report calls for enhanced supports for people living with mental health problems and illnesses to allow them to pursue education and obtain work. Strategic direction # 6 (CMHC, 2012) calls for strengthened human resources development. The corresponding recommendation for Action 6.2 and 6.3 seeks a pan-Canadian mental health workforce development strategy, including core competencies for all mental health service providers.

Competency has been defined as "a measurable capability that is required for effective performance" and is thought to be comprised of knowledge, skill and abilities and personal characteristics (Marelli, Tondora & Hoge 2005). There has been some evidence to suggest that the specific education of providers result in improved employment outcomes for clients they serve in public systems including higher employment rates and better wages after the attainment of provider degree (Van Houtte 2010).

The purpose of most certification efforts is to populate a profession with practitioners who are not only competent but also recognized as being competent to provide the unique services central to those fields. Leahy and Szymanski (1993), writing about the field of rehabilitation counseling, assert that one profession is distinguished from others when common structures are present, including self-regulation, autonomy, and monopoly. These common structures include programs of educational preparation, professional associations, accreditation of educational programs, regulation of practice, certification and licensing, and ethical mandates. From this assertion, it would seem that credentialing is essential to professionalize a field; yet many experts argue that credentialing is of questionable significance when little research exists supporting positive impact on the delivery of services.

Such is the case with the Psycho-social Vocational Rehabilitation [PVR] curriculum developed by Boston University. The curriculum is competency-based due to its level of clinical application and formal supervision of practice. However, this certificate program has been delivered over the past 10 years with no formal evaluation. The intent of this proposed research project is to evaluate the competency of the community mental health practitioners (e.g., social workers, occupational therapists, psychiatric nurses) enrolled in the PVR certificate program and the vocational outcomes of the clients they provide services to within their organization.

Linking practitioner competency in vocational rehabilitation to the improvement seen in their clients of attaining goals (CMHC, 2012) around employment and education has an opportunity to inform on how the community mental health workforce should be trained for the future for the benefit of their clients.

ELIGIBILITY:
Inclusion Criteria: any client who agreed to complete data collection form -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: clients with psychiatric disabilities utilizing vocational rehabilitation services in Winnipeg
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction with Vocational Services | 2 years
Practitioner perceived competency | 18 months

IPD SHARING:
Plan to Share IPD: No